CLINICAL TRIAL: NCT05163691
Title: A Phase 1 Study to Determine the Pharmacokinetics and Pharmacodynamics of Single and Multiple Inhaled Doses of GH001 in Healthy Volunteers
Brief Title: Pharmacokinetics of GH001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GH Research Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GH001-HV-103; 2021-000241-40 (EudraCT Number)
Record Dates: First submitted 2021-11-18; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: 5-MeO-DMT; 5-methoxy-N,N-dimethyltryptamine; 5-methoxy-dimethyltryptamine; Healthy Volunteers; Pharmacokinetics
MeSH Terms: interventions — Methoxydimethyltryptamines

STUDY DESIGN:
Intervention Model Description: This study will include separate single- and multiple-dose parts.
  Single-dose Part:
  A double-blind, placebo-controlled, randomized, parallel-group design with single, inhaled doses of GH001 in 3 groups of 10 subjects (randomized as 8 active and 2 placebo subjects per group):
  * Group A: single inhaled dose of 6 mg GH001
  * Group B: single inhaled dose of 12 mg GH001
  * Group C: single inhaled dose of 18 mg GH001
  Multiple-Dose Part:
  An open-label, non-randomized administration of up to 3 inhaled doses of GH001 within a single day (6 mg, followed by 12 mg, followed by 18 mg) with two different dose intervals (8 subjects per group):
  * Group D: 1-hour interval
  * Group E: 2-hour interval
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group A - 6 mg single-dose (Experimental): A single, inhaled dose of GH001 6 mg or placebo (randomized as 8 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Group B - 12 mg single-dose (Experimental): A single, inhaled dose of GH001 12 mg or placebo (randomized as 8 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Group C - 18 mg single-dose (Experimental): A single, inhaled dose of GH001 18 mg or placebo (randomized as 8 active and 2 placebo subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine; Drug: Placebo
- Group D - Individualized Dosing Regimen, 1-hour interval (Experimental): Administration of up to 3 inhaled doses of GH001 within a single day (6 mg, followed by 12 mg, followed by 18 mg) with a 1-hour dose interval (8 subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine
- Group E - Individualized Dosing Regimen, 2-hour interval (Experimental): Administration of up to 3 inhaled doses of GH001 within a single day (6 mg, followed by 12 mg, followed by 18 mg) with a 2-hour dose interval (8 subjects)
  Interventions: Drug: 5 Methoxy N,N Dimethyltryptamine

INTERVENTIONS:
Drug: 5 Methoxy N,N Dimethyltryptamine — GH001 administered via inhalation
  Other Names: GH001; 5-MeO-DMT
Drug: Placebo — GH001 Placebo administered via inhalation
  Other Names: GH001 Placebo
  Arms: Group A - 6 mg single-dose; Group B - 12 mg single-dose; Group C - 18 mg single-dose

SUMMARY:
The primary objective of this study is to investigate the serum pharmacokinetics of 5-MeO-DMT and its metabolite, bufotenine in healthy volunteers in a double-blind, placebo-controlled, randomized study design with single, inhaled doses of GH001 and in an open-label, non-randomized study design with intra-subject dose-escalation of GH001. As a secondary objective, the safety and tolerability of GH001, the mental health and well-being of the subjects after GH001 dosing(s), the pharmacodynamic profile of GH001 as evaluated by its psychoactive effects, and cognitive measures are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) in the range of 18.5 and 35.0 kg/m2 (inclusive);
* Subject is in good physical health in the opinion of the principal investigator (PI);
* Subject is in good mental health in the opinion of the PI and clinical psychologist;

Exclusion Criteria:

* Has known allergies or hypersensitivity or any other contraindication to 5-MeO-DMT;
* Has received any investigational medication within the last 4 weeks;
* Has a medical condition, which renders the subject unsuitable for the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-10-23 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic (PK) parameters derived from laboratory assay results of the systemic levels of 5-MeO-DMT and bufotenine | up to 4 hours
  For PK analyses, blood samples will be collected before and up to 4 hours after the administration of GH001 to determine 5-MeO-DMT and bufotenine serum concentrations.

SECONDARY OUTCOMES:
Safety: Adverse Event (AE) reporting | Up to 30 days
  Adverse events reported in the study and coded by MedDRA.
Safety: Frequency of clinically significant changes from baseline in electrocardiogram (ECG) recording | Up to 7 days
  Clinically significant changes in ECG include any significant change in rate or rhythm as determined by the principal investigator
Safety: Frequency of clinically significant changes from baseline in vital signs measurement | Up to 7 days
  Vital signs include heart rate (beats per minute), blood pressure (mmHg), respiratory rate (breaths per minute), oxygen saturation (%), and temperature (degrees celsius). Changes are defined as any clinically significant change from baseline as determined by the principal investigator
Safety: Frequency of clinically significant changes from baseline in safety laboratory tests of blood and urine | Up to 7 days
  Safety laboratory analyses are analyses of blood samples (biochemistry, hematology) and urine samples (urinalysis). Changes are defined as any clinically significant change from baseline as determined by the principal investigator.
Safety: Frequency of clinically significant changes from baseline in Peak Flow Respirometry | 1 hour after dosing
  Peak Flow is assessed using a standard peak flow respirometer, with the assessment done three times and the best of the three scores recorded as the final score (liters/minute).
Safety: Frequency of clinically significant changes from baseline in level of sedation | 30 minutes and 1 hour after dosing
  The Modified Observer's Assessment of Alertness and Sedation scale (MOAA/S) will be completed before and after GH001 dosing. Scored from 0 (deep sedation) to 5 (alert)
Safety: Change from baseline in Clinician Administered Dissociative States Scale (CADSS) | Up to 30 days
  Change from baseline in the Clinician Administered Dissociative States Scale (CADSS). The CADSS comprises 19 subjective items, ranging from 0 'not at all' to 4 'extremely. Summed together, these subscales form a total dissociative score. Combined score ranges from 0 to 76.
Safety: Assessment of Subject-Discharge readiness | up to 3 hours after last study drug administration
  Assessment of Discharge Readiness on the administration day by the Principal Investigator, using the Clinical Global Assessment of Discharge Readiness (CGADR).
Mental Health: Change from baseline in Brief Psychiatric Rating Scale (BPRS) | Up to 30 days
  Change from baseline in the Brief Psychiatric Rating Scale (BPRS). A scale to measure psychiatric symptoms. Each symptom is rated 1-7 and a total of 18 symptoms are scored. Combined score ranges from 18 to 126.
Mental Health: Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to 30 days
  Change from baseline in the Columbia-Suicide Severity Rating Scale (C-SSRS). A detailed questionnaire assessing both suicidal behaviour and suicidal ideation. No combined score is created.
Pharmacodynamic assessment: The dose-related psychoactive effects of GH001 as evaluated by a Visual Analogue Scale | up to 1 hour after dosing
  The Peak Experience Scale (PES) is a Visual Analogue Scale scored from 0-100
Pharmacodynamic assessment: 30-Question Mystical Experience Questionnaire (MEQ30) | up to 1 hour after dosing
  The MEQ30 is a validated procedure for assessing the extent of the psychoactive effects experienced by a subject. The validated MEQ30 uses thirty assessment questions across four areas of experience, all scored from 0 to 5.
Pharmacodynamic assessment: Challenging Experiences Questionnaire (CEQ) | up to 1 hour after dosing
  Completed by the subject after GH001 administration and assesses seven factors (grief, fear, death, insanity, isolation, physical distress, and paranoia) all scored from 0 to 5.
Pharmacodynamic assessment: Duration of the psychoactive effects (PsE) | up to 1 hour after dosing
  The duration of the experience, defined as time in minutes from drug administration to time when the subject reports that any psychoactive symptoms have subsided will be recorded.
Cognitive Function: Change from baseline in Psychomotor Vigilance Task (PVT) | Up to 7 days
  Change from baseline in the Psychomotor Vigilance Test (PVT). A computerized test assessing the reaction time in response to a visual stimulus. Outcome measures are Response Time and the number of attentional lapses (Response Time ≥ 500 msec).
Cognitive Function: Change from baseline in Auditory Verbal Learning Test (AVLT) | Up to 7 days
  The AVLT is one of the most widely used word learning tests in clinical research and practice. The test is based on successive auditory presentations of 15-word lists followed by attempted recall. The AVLT outcome measures are the rate of learning as well as the level of recall.
Cognitive Function: Change from baseline in Spatial Working Memory (SWM) task | Up to 7 days
  The SWM task requires retention and manipulation of visuo-spatial information. This self-ordered test provides a measure of strategy as well as working memory errors. The test involves a number of colored squares (boxes) shown on the screen which require a selection strategy to fill an empty column. The test takes about 4 minutes to complete. Outcome measures of the SWM include errors and strategy. The computerized Corsi Block will be the version of the SWM task used in this study.
Cognitive Function: Change from baseline in Digit Symbol Substitution Task (DSST) | Up to 7 days
  Change from baseline in the Digit Symbol Substitution Test (DSST). A computerized test with the task is to match digits with symbols from encoding list. The number of digits correctly encoded within 3 minutes is the performance measure.

CONTACTS AND LOCATIONS:
Overall Officials: GH Research Clinical Team, Study Director — GH Research Ireland Limited
Locations (1):
- GH Research Clinical Trial Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GH Research Company Website — http://www.ghres.com